CLINICAL TRIAL: NCT01941784
Title: Taking Health Realization Into Valued Eating and Exercise (THRIVE): A Feasibility Study of an Intervention to Prevent Weight Gain for Breast Cancer Survivors During Chemotherapy
Brief Title: Health Education Intervention in Reducing Weight Gain in Patients With Newly Diagnosed Stage I-IV Breast Cancer Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00025131; NCI-2013-01742 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 97513 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2018-07

CONDITIONS: Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Early Intervention, Educational; Methods; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (health education program) (Experimental): See Detailed Description.
  Interventions: Other: educational intervention; Other: counseling intervention; Behavioral: telephone-based intervention; Other: questionnaire administration; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: educational intervention — Undergo health education program
  Other Names: intervention, educational
Other: counseling intervention — Undergo health education program
  Other Names: counseling and communications studies
Behavioral: telephone-based intervention — Receive follow-up phone calls
Other: questionnaire administration — Ancillary studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This pilot clinical trial studies a health education intervention in reducing weight gain in patients with newly diagnosed stage I-IV breast cancer undergoing chemotherapy. A health education program may reduce weight gain and improve quality of life in patients undergoing chemotherapy for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of conducting a weight maintenance intervention, in terms of recruiting and retaining participants.

II. To obtain preliminary data on the effectiveness of an intervention to prevent weight gain on body composition, self-efficacy, perceived stress, fatigue, depression, exercise capacity, and health-related quality of life (HRQL). Changes in physical activity and dietary intake will also be monitored.

III. To determine if the weight control protocol requires refinement for use in a randomized controlled trial.

IV. To determine how many participants opt to enroll in a short-term healthy lifestyle program at completion of the final testing visit.

OUTLINE:

Participants undergo four 30-60 minute health education sessions and 3 follow-up phone sessions with an interventionist trained in behavioral science, physical activity and nutrition, and positive psychology over 12 months.

EDUCATION SESSION I: Participants receive information from the interventionist concerning healthy diet choices and exercise and begin to keep a food log.

EDUCATION SESSION II: Interventionists review information from session I and patient food logs. Participants receive recommendations for exercise and set activity goals.

EDUCATION SESSION III: Participants receive information on how to determine portion sizes and the importance of strength training and building lean muscle mass.

EDUCATION SESSION IV: Interventionists review information from the previous 3 sessions and discuss the importance of planning and goal setting with participants. The interventionist also discusses physical and mental barriers to exercise.

After completion of the education sessions, patients receive 3 phone calls at times convenient to the patient to answer questions about information learned in previous educational sessions.

After completion of study, participants are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Women with newly-diagnosed breast cancer, stage I-IV who are within first two rounds of chemotherapy
* 3.1.2 Women who are receiving, or scheduled to receive, one of the following classes of therapy in the adjuvant or neo-adjuvant setting: anthracyclines, taxanes, cyclophosphamide, or trastuzumab. Participants must be within their first two rounds of chemotherapy - Body mass index (BMI) > 20
* Treating physician approval to participate in study
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document

Exclusion Criteria:

* Diagnosis of recurrent breast cancer
* Women who are already participating in a formal or medically prescribed weight management program
* Women who have already completed more than two rounds of chemotherapy
* Women who are pregnant or nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-11-25 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-04-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of conducting the weight gain prevention intervention, measured as the percent of screened participants that are eligible and agree to participate | Baseline
  Reasons why participants are not eligible will be reported and inclusion/exclusion criteria will be reevaluated. The proportion of participants who completed all sessions and testing visits will be estimated and compared. Barriers to recruitment (e.g., timing of intervention, inconvenience, time constraints, participant feeling too sick) will be recorded to assist in designing the larger trial.

SECONDARY OUTCOMES:
Effect of the intervention on body composition | Up to 52 weeks
  Descriptive statistics consisting of frequency tables and percents for categorical variables and means, medians, standard deviations, and ranges for continuous variables will be tabulated. Repeated-measure analysis of covariance (ANCOVAs) to test for change in our primary variables over the 3 timepoints will be conducted, controlling for baseline differences. Additionally, effect sizes will be calculated as they account for sample size and are useful when a lack of power leads to nonsignificant findings. These estimates of variability will be used when designing a future trial.
Effect of the intervention on self-efficacy | Up to 52 weeks
  Descriptive statistics consisting of frequency tables and percents for categorical variables and means, medians, standard deviations, and ranges for continuous variables will be tabulated. Repeated-measure ANCOVAs to test for change in our primary variables over the 3 timepoints will be conducted, controlling for baseline differences. Additionally, effect sizes will be calculated as they account for sample size and are useful when a lack of power leads to nonsignificant findings. These estimates of variability will be used when designing a future trial.
Effect of the intervention on perceived stress | Up to 52 weeks
  Descriptive statistics consisting of frequency tables and percents for categorical variables and means, medians, standard deviations, and ranges for continuous variables will be tabulated. Repeated-measure ANCOVAs to test for change in our primary variables over the 3 timepoints will be conducted, controlling for baseline differences. Additionally, effect sizes will be calculated as they account for sample size and are useful when a lack of power leads to nonsignificant findings. These estimates of variability will be used when designing a future trial.
Effect of the intervention on fatigue | Up to 52 weeks
  Descriptive statistics consisting of frequency tables and percents for categorical variables and means, medians, standard deviations, and ranges for continuous variables will be tabulated. Repeated-measure ANCOVAs to test for change in our primary variables over the 3 timepoints will be conducted, controlling for baseline differences. Additionally, effect sizes will be calculated as they account for sample size and are useful when a lack of power leads to nonsignificant findings. These estimates of variability will be used when designing a future trial.
Effect of the intervention on 6 minute walk distance | Up to 52 weeks
  Descriptive statistics consisting of frequency tables and percents for categorical variables and means, medians, standard deviations, and ranges for continuous variables will be tabulated. Repeated-measure ANCOVAs to test for change in our primary variables over the 3 timepoints will be conducted, controlling for baseline differences. Additionally, effect sizes will be calculated as they account for sample size and are useful when a lack of power leads to nonsignificant findings. These estimates of variability will be used when designing a future trial.
Effect of the intervention on fruit, vegetable, and fat intake | Up to 52 weeks
  Descriptive statistics consisting of frequency tables and percents for categorical variables and means, medians, standard deviations, and ranges for continuous variables will be tabulated. Repeated-measure ANCOVAs to test for change in our primary variables over the 3 timepoints will be conducted, controlling for baseline differences. Additionally, effect sizes will be calculated as they account for sample size and are useful when a lack of power leads to nonsignificant findings. These estimates of variability will be used when designing a future trial.
Effect of the intervention on physical activity participation | Up to 52 weeks
  Descriptive statistics consisting of frequency tables and percents for categorical variables and means, medians, standard deviations, and ranges for continuous variables will be tabulated. Repeated-measure ANCOVAs to test for change in our primary variables over the 3 timepoints will be conducted, controlling for baseline differences. Additionally, effect sizes will be calculated as they account for sample size and are useful when a lack of power leads to nonsignificant findings. These estimates of variability will be used when designing a future trial.
Effect of the intervention on health-related quality of life | Up to 52 weeks
  Descriptive statistics consisting of frequency tables and percents for categorical variables and means, medians, standard deviations, and ranges for continuous variables will be tabulated. Repeated-measure ANCOVAs to test for change in our primary variables over the 3 timepoints will be conducted, controlling for baseline differences. Additionally, effect sizes will be calculated as they account for sample size and are useful when a lack of power leads to nonsignificant findings. These estimates of variability will be used when designing a future trial.
Sample size for future larger trials | Up to 52 weeks
  Data from outcomes 1 and 2 along with qualitative data, will allow researchers to refine the protocol accordingly.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Mihalko, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States